CLINICAL TRIAL: NCT05563376
Title: Prospektive Erfassung Von standardmäßig Erhobenen Daten im Rahmen Der Erlanger Fontan-Sprechstunde Zur Behandlung Und Überwachung Von PatientInnen Mit univentrikulärem Herzfehler im Sinne Einer Fontan-Zirkulation
Brief Title: Fontan-Sprechstunde
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21-195_1-B
Record Dates: First submitted 2022-09-21; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Univentricular Heart
MeSH Terms: conditions — Univentricular Heart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCPC completed (Other): All patients after TCPC completion
  Interventions: Diagnostic Test: Univentricular Hearts

INTERVENTIONS:
Diagnostic Test: Univentricular Hearts — Prevention when factors are recognized

SUMMARY:
After successful Fontan surgery, the risk of mortality in childhood is only low. Unfortunately, some of the patients suffer from Fontan-typical long-term complications in the long-term course, whereby protein loss neuropathy must be mentioned in particular, which is described in the literature with an incidence of 3-14% (1, 2) and still has a 5-year risk of death of 6-12% today (2, 3). Protein loss tereopathy leads to loss of protein in the intestine and subsequently to diarrhea and edema. Other problems concern the liver, which can develop cirrhosis due to chronic congestion (4-6). Cardiac can lead to heart failure and arrhythmias.

The registry study described in this protocol is intended to identify factors that influence the treatment outcome of patients in the Fontan circulation in the long term through systematic prospective documentation of the data from our standardized and guideline-oriented treatment.

DETAILED DESCRIPTION:
In particular, the following points will be scientifically analyzed:

1. The development of lymphatic drainage disorders (7-9)
2. The cellular changes of the immunological system and metabolome (10) In addition to the clinical routine, weight-adapted EDTA blood for the isolation of peripheral blood mononuclear cells (PBMCs) for the scientific investigation of immunological changes and serum for the analysis of the metabolome will be examined at three times (Figure 1: Times 2, 4, 7) as part of a routine blood sample (10).
3. The recording and treatment of psychological, social and developmental abnormalities with the help of standardized questionnaires.
4. The evaluation of special sonography examinations of the liver and kidney in the long-term course, as well as their treatment.
5. The assessment of the hemodynamic peculiarities and the classification with regard to Cardiac function in the long-term course of patients with Fontan circulation.
6. The assessment of various laboratory parameters as risk parameters for the development of complications.
7. The recording of cardiopulmonary performance in the long-term course and its ability to be influenced by education regarding sporting activity and the handing over of an individualized training plan.
8. The influence of physical activity on possible complications of Fontan circulation.
9. The influence of early psychological, nutritional, or social intervention in the event of abnormalities on later complications of Fontan circulation.

ELIGIBILITY:
Inclusion Criteria:

* congenital heart defect of the univentricular type that has led to Fontan circulation

Exclusion Criteria:

* no exclusion criteria

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2031-09-01 (Estimated); Study Completion 2041-09-01 (Estimated)

PRIMARY OUTCOMES:
Reducing mortality and morbidity and improving quality of life in long-term care for Fontan patients | 50 Jahre
  1. Fontan Tunnel Obstruction
  2. Fontan-typical klin. Symp. defined in points 5.+6. o. Presence of edema, ascites, susceptibility to infections, reduced resilience, cyanosis, lack of size and weight development, diarrhea
  3. Heart or heart valve insufficiency defined as end-diastolic volume/BSA (EDP corrected) above the norm, ventricle ejection fraction (EF) <50%, atrioventricular heart valve insufficiency (AVI) >grade 2, aortic valve insufficiency >grade 2
  4. Pathological lymphatic vessel imaging defined as lymphatic vasodilation (LAE) type ≥ 3 according to Biko et al. (abnormal supraclavicular lymphatic vasodilation with infiltration of the mediastinum) (7). Presence of mesenteric lymphatic vascular congestion (8)
  5. Hypoproteinaemia defined as serum albumin <3.4 mg/dl (4), total protein (TP) <50 g/l
  6. protein-losing enteropathy (PLE) defined as (3, 4)
  7. Failing Fontan defined as Operative Fontan Take-down, Listing for Heart Transplantation and/or Death

CONTACTS AND LOCATIONS:
Overall Officials: Sven Dittrich, Prof., Study Chair — Universitätsklinikum Erlangen
Locations (1):
- Universitätsklinikum, Erlangen, Germany